CLINICAL TRIAL: NCT04697654
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Inhaled TLC19 in Healthy Volunteers
Brief Title: The Safety, Tolerability, and Pharmacokinetics of Inhaled TLC19 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TLC19A1001
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-09

CONDITIONS: COVID-19
Keywords: hydroxychloroquine; Inhalation
MeSH Terms: conditions — COVID-19; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- TLC19 (low dose) (Experimental): TLC19 2ml single dose
  Interventions: Drug: TLC19
- TLC19 (medium dose) (Experimental): TLC19 4ml single dose
  Interventions: Drug: TLC19
- TLC19 (high dose) (Experimental): TLC19 6ml single dose
  Interventions: Drug: TLC19
- TLC19 Vehicle (low dose) (Sham Comparator): TLC19 Vehicle 2ml single dose
  Interventions: Drug: TLC19 Vehicle
- TLC19 Vehicle (medium dose) (Sham Comparator): TLC19 Vehicle 4ml single dose
  Interventions: Drug: TLC19 Vehicle
- TLC19 Vehicle (high dose) (Sham Comparator): TLC19 Vehicle 6ml single dose
  Interventions: Drug: TLC19 Vehicle

INTERVENTIONS:
Drug: TLC19 — Hydroxychloroquine Liposome Inhalation Suspension
  Other Names: TLC19 (Hydroxychloroquine Liposome Inhalation Suspension)
  Arms: TLC19 (high dose); TLC19 (low dose); TLC19 (medium dose)
Drug: TLC19 Vehicle — Liposome Inhalation Suspension (same formulation as TLC19 but without the active ingredient, HCQ)
  Other Names: TLC19 Vehicle (same formulation as TLC19 but without the active ingredient)
  Arms: TLC19 Vehicle (high dose); TLC19 Vehicle (low dose); TLC19 Vehicle (medium dose)

SUMMARY:
Phase 1 randomized, vehicle-controlled, blinded study to assess the safety, tolerability, and PK of single ascending doses of inhaled TLC19 in healthy volunteer subjects.

DETAILED DESCRIPTION:
A Phase 1 randomized, vehicle-controlled, blinded study to assess the safety, tolerability, and PK of single ascending doses of inhaled TLC19 (Hydroxychloroquine Liposome Inhalation Suspension) in healthy volunteer subjects. Three dose levels will be assessed in sequential cohorts, with 2 mL, 4 mL, and 6 mL. Total of approximately 30 subjects will be randomized in the study in 3 cohorts. Subjects will be enrolled and randomized to receiving either TLC19 or TLC 19 Vehicle.

Drug Administration: Blinded study medication will be administered through inhalation via a portable vibration mesh nebulizer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 65 years of age
2. Body mass index (BMI) 18.0 to 30.0 kg/m2.
3. Never-smoker

Exclusion Criteria:

1. Body weight <50 kg
2. Donation of blood (450 mL) or blood loss within 3 months prior to study
3. Contraindication, allergy, or hypersensitivity to hydroxychloroquine or chloroquine or other 4 aminoquinolines
4. Use of any prescription or OTC medications or herbal supplements within 2 weeks (or 5half-lives if longer) prior to study
5. Use of any investigational product/medical device within 30 days or 5 half-lives prior to study, or participation in ≥4 investigational drug studies within 1 year prior to study
6. History or presence of any of the following conditions:

   * Autoimmune or rheumatoid inflammatory disease
   * Cardiac disorders
   * Lung disease, prior intubation, or requiring use of an inhaler
   * Liver cirrhosis or Child-Pugh class C
   * Retinopathy or maculopathy
   * Neuromuscular diseases
   * Glucose-6 phosphate dehydrogenase deficiency
   * Hematologic malignancy
   * Chronic kidney disease or renal failure
   * Psoriasis or porphyria
   * Diabetes mellitus
   * Severe allergic or anaphylactic reactions
   * Any other significant condition that would preclude participation
7. History of substance abuse or dependency in the last 12 months, or a history of recreational intravenous drug use over the last 5 years
8. Fever or symptomatic viral or bacterial infection within 2 weeks prior to study
9. Any clinically significant laboratory abnormality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs | 0-28 Days
  To evaluate the severity, seriousness, outcome, and action taken of AE

SECONDARY OUTCOMES:
Maximum blood concentration | 0-168 hours
  Cmax
Time to reach maximum blood concentration | 0-168 hours
  Tmax
Area under the blood concentration-time curve | 0-168 hours
  AUC0-last

CONTACTS AND LOCATIONS:
Overall Officials: Carl Brown, PhD, Study Director — Taiwan Liposome Company, Ltd.
Locations (1):
- Mackay Memorial Hospital Tamsui Branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No